CLINICAL TRIAL: NCT03018457
Title: Evaluation of Trabecular Microarchitecture of the Alveolar Bone by Micro-computed Tomography and of Osseointegration of Dental Implants by Resonance Frequency Analysis: Correlation Study.
Brief Title: Evaluation of Trabecular Microarchitecture of the Alveolar Bone by Micro-computed Tomography and of Osseointegration of Dental Implants by Resonance Frequency Analysis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608111; ANSM (Other: 2016-A01680-51)
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-02

CONDITIONS: Dental Implant
Keywords: Trabecular microarchitecture; alveolar bone; osseointegration; dental implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients who need a dental implants
  Interventions: Device: ISQ

INTERVENTIONS:
Device: ISQ — Measured by Osstell.

SUMMARY:
Dental implants are a prosthetic rehabilitation device whose success depends of the bone morphology and quality, in more the surgical procedure.

This study aims to assess whether the parameters of the trabecular microarchitecture of alveolar bone taken from the site of the placement of the dental implant, calculated by micro-CT are correlated with ISQ (implant stability quotient) using the Osstell according the principle of the resonance frequency analysis at the 10th postoperative week during the osseointegration of dental implants (secondary stability).

The cortical alveolar bone is a recognized factor in the phase of primary stability of osseointegration. The role of trabecular bone in the secondary stability is not clearly determined.

DETAILED DESCRIPTION:
The aim of this study is to check whether the trabecular bone with its microarchitecture plays a predictive role in osseointegration of dental implants precisely in its biological stability phase or its secondary stability phase.

If this correlation is established, a larger study must be conducted to identify a profile of patients at risk for failure of osseointegration of the dental implant.

ELIGIBILITY:
Inclusion Criteria:

* affiliated patient or entitled to a social security scheme
* requiring the installation of one or more dental implants
* partial or total loss teeth, the height and width od the alveolar bone does not require bone grafting or guides regeneration

Exclusion Criteria:

* patient who underwent pre-implant surgery (bone grafting, elevation of the maxillary sinus, guided regeneration)
* patient under corticosteroid therapy in the long term
* patient who benefited from the head and neck radiotherapy
* patient under bisphosphonates intravenously treatment
* all cases immediate implantation and extraction of all implant put into immediate expenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need a dental implant
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) | 10 weeks
  The Osstell is a portable hand instrument used to measure the stability of the dental implant according to the principle of the resonance frequency analysis. It is allow to measure the ISQ.

SECONDARY OUTCOMES:
volume fraction of the bone | 10 weeks
  Measured by Scanco microscanner
thickness between trabecular | 10 weeks
  Measured by Scanco microscanner
Thickness of trabecular | 10 weeks
  Measured by Scanco microscanner
trabecular separation | 10 weeks
  Measured by Scanco microscanner
trabecular number | 10 weeks
  Measured by Scanco microscanner
structural model index | 10 weeks
  Measured by Scanco microscanner
trabecular pattern factor | 10 weeks
  Measured by Scanco microscanner
connectivity density | 10 weeks
  Measured by Scanco microscanner
degree of anisotropy | 10 weeks
  Measured by Scanco microscanner

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Cabinet dentaire MOLIMARD, Le Puy-en-Velay, France

IPD SHARING:
Plan to Share IPD: No